CLINICAL TRIAL: NCT04123691
Title: Cardio-respiratory Events in VLBW Preterm Infants During the Transitional Period: Clinical Features and Impact of Neonatal Characteristics.
Brief Title: Cardio-respiratory Events in Preterm Infants During Transition
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Silvia Martini, PhD student, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-CRE-1
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Apnea of Prematurity; Apneic Spells of Newborn Nos; Patent Ductus Arteriosus; Premature Birth; Desaturation of Blood; Bradycardia Neonatal
Keywords: cardio-respiratory events; preterm infants; transitional period; desaturation; bradycardia; apnea
MeSH Terms: conditions — Apnea; Ductus Arteriosus, Patent; Premature Birth; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: pulse oximetry monitoring — pulse oximetry monitoring as per routine clinical practice

SUMMARY:
Cardio-respiratory events (CRE), defined as intermittent episodes of hypoxemia and/or bradycardia, are particularly common among preterm infants. It has been previously shown that CRE result in transient brain hypoxia and hypoperfusion and may represent a possible risk factor for neurodevelopmental impairment and retinopathy of prematurity. The high cardio-respiratory instability typically seen in preterm infants during the first 72 hours of life may influence CRE occurrence, with possible clinical implications. This study aims to characterize CRE features in this transitional period and to evaluate whether specific neonatal and clinical characteristics are associated with different CRE types.

Newborn infants with gestational age (GA) <32 weeks or birth weight (BW) <1500 g are enrolled. Congenital malformations and mechanical ventilation are exclusion criteria. During the first 72 hours, heart rate (HR) and peripheral oxygen saturation (SpO2) are continuously monitored, and an echocardiogram is performed to assess the status of the ductus arteriosus. CRE are clustered into isolated desaturation (ID, SpO2<85%), isolated bradycardia (IB, HR<100 bpm or <70% baseline), combined desaturation and bradycardia (DB, occurrence of the two events within a 60-sec window). According to their duration and SpO2 and/or HR nadir values, CRE are also classified as mild (SpO2 80-84% and HR 80-100 bpm and duration <60 sec), moderate (SpO2 70-79% or HR 80-60 bpm or duration 61-120 sec) or severe (SpO2 <70% or HR <60 bpm or duration >120 sec). A generalized estimating equation (GEE) will be used to examine the impact of relevant variables on CRE type and severity.

DETAILED DESCRIPTION:
Background Cardio-respiratory events (CRE), defined as intermittent hypoxic and/or bradycardic episodes, are very common among premature infants. The poor respiratory drive, together with the increased metabolic oxygen consumption and the reduced total blood oxygen carrying capacity of this population significantly enhance CRE frequency and severity.

Evidence from animal models has shown that CRE, either alone or combined to specific clinical factors (i.e., intrauterine growth restriction, support modality, need for supplemental oxygen etc.), can trigger oxidative stress, which may contribute to adverse neonatal outcomes. In particular, a significant association between CRE and the development of retinopathy of prematurity (ROP) has been largely established, with evidence of a positive correlation between ROP severity and CRE duration, depth of desaturation, and persistency after 3 to 5 weeks of age. A critical role for CRE on early brain development has also been suggested by several studies showing a relationship between the ensuing hypoxic burden and poor neurodevelopment from early infancy up to early school age. Eventually, a possible association between CRE severity and the development of bronchopulmonary dysplasia has been recently reported in very-low-birth-weight (VLBW) neonates.

Most of the available literature on CRE characteristics, physiological mechanisms and effects in the premature population, however, is based on infants aged 2-weeks or older, while data from the transitional period, defined as the first 72 hours after birth, are scarce.

The transitional period represents a critical phase of physiological adaptation and may affect several organ systems, most notably the heart and the lungs. In particular, the dynamic cardiovascular changes that characterize the transition from fetal to neonatal circulation may enhance preterm infants' cardiorespiratory instability, with possible effects on CRE characteristics. In turn, the hemodynamic and respiratory disturbances that characterize post-natal transition may exacerbate the clinical burden of CRE during this period, with possible clinical implications.

This study aims to characterize CRE during transitional periods in VLBW preterm infants, and to evaluate whether specific neonatal characteristics may have an influence on CRE type and severity.

Methods Infants born at S. Orsola-Malpighi Hospital are consecutively enrolled in this observational, prospective study if fulfilling the following eligibility criteria: gestational age (GA) <32 weeks' gestation, birth weight <1500 g, 0-12 hours of life, written informed consent obtained from the parents/legal guardians of each infant.

Peripheral oxygen saturation (SpO2) and heart rate (HR) are routinely monitored during hospital stay using a Masimo Radical 7 (Masimo Corporation, Irvine, CA, USA) pulse oximeter with a 1-Hz sampling frequency.

Isolated desaturations (ID) are defined as SpO2 <85% and classified into mild (SpO2 80-84%), moderate (SpO2 70-79%) and severe (SpO2 <70%).

Isolated bradycardias (IB) are defined as any HR drop <100 bpm or >30% from baseline values, calculated daily over the first 72 hours of life, and further stratified into mild (HR 80-100 bpm or any drop between 31-50% of the baseline), moderate (HR 60-79 bpm or any drop between 51-70% of baseline) or severe (HR <60 bpm or any drop >70% of baseline).

Desaturations and bradycardias occurring within a 60-sec time window are considered as combined events (DB).

Event duration is calculated as the period spent below the SpO2 and HR thresholds described for CRE definition. According to their duration, CRE are defined as mild (10-60 sec), moderate (61-120 sec), or severe (>120 sec).

Neonatal clinical characteristics The following antenatal and neonatal data are tracked down on a specific case report form: GA, antenatal steroids (complete course vs. incomplete course or not given) evidence of reversed end-diastolic flow at antenatal umbilical Doppler (uREDF) (present vs. absent); ventilatory status over the first 72 hours of life (continuous positive airway pressure [CPAP] vs. nasal cannulas or self-ventilating in air [SVIA]).

A screening echocardiogram is routinely performed at the time of enrollment using an ultrasound scanner CX50 (Philips Healthcare) with a 12-MHz probe, and repeated 6-12 hourly in the presence of a patent ductus arteriosus (PDA) or 12-24 hourly if there is no evidence of PDA. Based on echocardiographic features, the ductal status is classified as follows: no evidence of PDA (noPDA), restrictive PDA (rPDA; restrictive shunt pattern and left atrium to aortic root ratio [LA:Ao] ratio <1.5), hemodynamically significant PDA (hsPDA; pulsatile shunt pattern, LA:Ao ratio ≥1.5 or presence of reversed end-diastolic flow (REDF) either in the descending aorta or in the anterior cerebral artery).

Statistical analysis Generalized estimating equation (GEE) models will be used to analyze the effect of GA, uREDF, antenatal steroids, ductal and ventilatory status on CRE type (ID, IB, DB) and severity (mild, moderate and severe) and the relation of different neonatal characteristics and event types with event duration. Variations in the daily number of ID, IB and DB over the 3 days of life, adjusted for the effective hours of recording, will be analyzed using Repeated Measures ANOVA (RM-ANOVA). IBM SPSS, version 25.0, will be used for statistical analysis. The significance level is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

- gestational age <32 weeks and/or birth weight <1500 g

Exclusion Criteria:

* mechanical ventilation
* major congenital malformations
* genetic abnormalities

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm newborns age 0 to 72 hours of life with non-invasive ventilatory support.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Definition of CRE characteristics | 0-72 hours of life
  Total number of desaturations, bradycardias and combined events
Time distribution of CRE | 0-72 hours of life
  Daily incidence of desaturations, bradycardias and combined events
Effect of neonatal characteristics on CRE type | 0-72 hours of life
  Generalized estimating equation (GEE) analysis evaluating the effect of GA, uREDF, antenatal steroids, ductal and ventilatory status on CRE type (ID, IB, DB) using multinomial distribution/probit link.
Effect of neonatal characteristics on CRE severity | 0-72 hours of life
  Generalized estimating equation (GEE) analysis evaluating the effect of GA, uREDF, antenatal steroids, ductal and ventilatory status on CRE severity (mild, moderate and severe) using multinomial distribution/probit link.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Martini, MD, Principal Investigator — Sant'Orsola-Malpighi University Hospital, Bologna, Italy
Locations (1):
- Sant'Orsola-Malpighi University Hospital, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No